CLINICAL TRIAL: NCT01466270
Title: A Feasibility Study of Donepezil in Female Breast Cancer Survivors With Self-Reported Cognitive Dysfunction Following Chemotherapy
Brief Title: Study of Donepezil in Female Breast Cancer Survivors With Cognitive Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00019792-1; U10CA081851 (NIH); REBACCCWFU 97211 (Other: NCI)
Record Dates: First submitted 2011-11-02; First posted 2011-11-07 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Anxiety Disorder; Breast Cancer; Cognition Disorders; Depression; Fatigue; Sleep Disorders
Keywords: fatigue; sleep disorders; depression; anxiety disorder; cognitive/functional effects; breast cancer; cancer survivor
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Cognition Disorders; Depression; Fatigue; Sleep Wake Disorders | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (Experimental): Patients receive donepezil hydrochloride PO QD.
  Interventions: Drug: donepezil hydrochloride
- Arm II (Placebo Comparator): Patients receive placebo PO QD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: donepezil hydrochloride — Given PO
  Other Names: Donepezil
  Arms: Arm I
Drug: Placebo — Given PO
  Arms: Arm II

SUMMARY:
RATIONALE: Donepezil hydrochloride may help lessen cognitive dysfunction caused by chemotherapy.

PURPOSE: This phase II trial is studying donepezil hydrochloride in treating cognitive dysfunction after chemotherapy in female breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of conducting a randomized placebo-controlled clinical trial for cognitive symptoms in female breast cancer survivors.

Secondary

* Estimate the variability of the clinical outcomes (FACT-Cognition Perceived Cognitive Impairment subscale, neurocognitive battery, FACIT-Fatigue, FACT Cog Total Score, PROMIS Fatigue, Epworth Sleepiness Scale, Beck Depression Inventory, Beck Anxiety Inventory, and RAND Short Form-36).
* Estimate the within patient correlation over time of the clinical outcomes.
* Obtain preliminary estimates of the effect of donepezil on the primary and secondary outcome variables.
* Correlate the reports of fatigue, sleep disturbance, and mood with measures of cognitive symptoms and neurocognitive test performance.
* Document the severity of cognitive symptoms and functional impairment in female breast cancer survivors who enroll on this pilot study.
* Correlate cognitive symptoms with cognitive test performance.
* Document the toxicities associated with donepezil hydrochloride use.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to menopausal status (pre- vs peri-/post-menopausal) and time since end of chemotherapy (12-36 months vs 36.01-60 months).

Arm I: Patients receive donepezil hydrochloride orally (PO) once daily (QD).

Arm II: Patients receive placebo PO QD.

In both arms treatment continues for 24 weeks.

Patients complete the entire battery of neurocognitive tests and questionnaires (FACT-Cognition Perceived Cognitive Impairment subscale, neurocognitive battery, FACIT-Fatigue, FACT Cog Total Score, PROMIS Fatigue, Epworth Sleepiness Scale, Beck Depression Inventory, Beck Anxiety Inventory, and RAND Short Form-36) at baseline (pre-treatment), 24 weeks (end of medication), and 36 weeks (end of wash-out).

After completion of therapy, patients are followed at 12 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

* Adults >18 years old.
* Female with history of invasive breast cancer
* Must have completed adjuvant chemotherapy between 1 and 5 years prior to registration
* Received at least 4 cycles of cytotoxic chemotherapy
* Documentation of prior chemotherapy
* Patients receiving ongoing hormonal therapy for breast cancer must be on the same hormonal agent for at least 3 months prior to study registration and continue for the duration of the study (9 months)
* Karnofsky Performance Status must be > 60 or ECOG 0-2.
* Use of psychotropic medications (anti-depressants, anxiolytics, sleeping aids, narcotics) is permitted. Patient will be asked to list any that have been taken within the last 3 days on the recent medication sheet.
* Patients must be able to give informed consent to participate in the study, including signing the consent form.
* Self-reported cognitive disruption (FACT-Cog Version 3 Perceived Cognitive Impairments sub-score of < 63)
* Negative serum pregnancy test within 10 days prior to registration for women of child-bearing potential.

EXCLUSION CRITERIA:

* Evidence or suspected recurrent or metastatic disease
* History of dementia, Alzheimer's disease, multi-infarct dementia or CVA (history of transient ischemic attack (TIA is allowed)
* Current use of donepezil, galantamine, rivastigmine, tacrine, memantine, methylphenidate, dextroamphetamine, or any other specific cognition enhancing drugs.are not allowed. For patients who have used these medications they must not have used them within 4 weeks prior to registration.

Patients may not currently be taking Ketoconazole or Quinidine

* Hypersensitivity to donepezil.
* Use of investigational medications within the last 30 days.
* Prior brain metastasis
* Traumatic brain injury, multiple sclerosis or recent myocardial infarction
* History of schizophrenia, psychosis or substance abuse
* Untreated current severe depression. (Currently treated depression is permitted if treatment is stable.)
* Acute severe fatigue, chronic fatigue syndrome or fibromyalgia.
* History of hepatic or renal dysfunction or disease
* Pregnant women are excluded from this study. The effects of donepezil on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because donepezil is known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* It is unknown whether donepezil is excreted in breast milk, for this reason women who are currently breast-feeding are not eligible for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia A. Lawrence, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were accrued between 7/12 and 1/13 from CCOP sites across the nation.
Pre-assignment Details: No wash-out or run-in period. All enrolled patients were randomized.
Groups:
- Arm I - Donepezil: Patients receive donepezil hydrochloride PO QD.
- Arm II - Placebo: Patients receive placebo PO QD.
Period: Overall Study
Arm/Group | Arm I - Donepezil | Arm II - Placebo
Started | 31 | 31
Completed | 19 | 25
Not Completed | 12 | 6
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 3
Not completed — Progression | 1 | 0
Not completed — Toxicity | 4 | 1
Not completed — Multiple | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Donepezil | Arm II - Placebo | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 27 | 51
  >=65 years | 7 | 4 | 11
Age, Continuous [Median (Full Range); unit: years] | 56 [39 to 79] | 56 [41 to 78] | 56 [39 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 27 | 29 | 56
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Retention is the percentage of participants who stay in the study for 24 weeks.
Time Frame: 24 Weeks
Population: All randomized patients
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 31 | 31
percentage of participants | 71.0 (8.3) | 80.7 (7.2)

2. Primary Outcome: Compliance
Description: Compliance is the percentage of pills taken while on study (based on returned diaries)
Time Frame: 24 weeks
Population: Participants who returned pill diaries. Note that some participants did not return diaries so the numbers of participants for this analysis may not agree with the numbers for other analyses.
Measure: Mean (Full Range); unit: percentage of pills
Arm/Group | Arm I - Donepezil | Arm II - Placebo
Number analyzed (Participants) | 26 | 27
percentage of pills | 98.0 [89.6 to 100.0] | 98.0 [89.6 to 100.0]

3. Secondary Outcome: HVLT-IR
Description: Hopkins verbal learning test - immediate recall is the number of words (of 12) than can be remembers during three tries. The total score ranges from 0 to 36. Higher is better.
Time Frame: 24 weeks
Population: All randomized participants except two who did not provide any data.
Measure: Least Squares Mean (Standard Error); unit: number of words recalled
Arm/Group | Arm I - Donepezil | Arm II - Placebo
Number analyzed (Participants) | 30 | 30
number of words recalled | 25.58 (1.36) | 22.94 (1.24)

4. Secondary Outcome: Fatigue
Description: Fatigue is quantified by the FACIT-Fatigue scale. It consists of 13 questions answered on a 0 to 4 point scale. The fatigue score is the sum of the responses (some reverse scored) so that higher values represent less fatigue.
Time Frame: 24 weeks
Population: All randomized participants except two who did not provide any data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Donepezil | Arm II - Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 35.89 (2.20) | 35.51 (2.02)

ADVERSE EVENTS:
Time Frame: 40 weeks (one month following the end of the study)
Description: The numbers of participants for this analysis may not agree with the numbers for the other analyses as not all participants completed their AE/toxicity evaluations.
Arm/Group | Arm I - Donepezil | Arm II - Placebo
Serious Adverse Events (participants affected / at risk) | 2/28 | 1/30
Other Adverse Events (participants affected / at risk) | 28/28 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Donepezil (N=28) | Arm II - Placebo (N=30)
Insomnia (General disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain: Chest Wall (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Donepezil (N=28) | Arm II - Placebo (N=30)
Anorexia (General disorders) | 4 (5) | 7 (11)
Cognitive Disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (11) | 6 (9)
Fatigue (General disorders) | 20 (49) | 19 (49)
Headache (Nervous system disorders) | 11 (15) | 8 (15)
Insomnia (General disorders) | 18 (37) | 21 (49)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 15 (29) | 8 (14)
Nausea (Gastrointestinal disorders) | 8 (10) | 8 (12)
Neuropathy: sensory (Nervous system disorders) | 3 (5) | 2 (3)
Pain: joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes